CLINICAL TRIAL: NCT04615481
Title: Effects of Elliptical Training Versus Ergo-meter on Cardiopulmonary Parameters in Post CABG Patients
Brief Title: Elliptical Training Versus Ergo-meter on Cardiopulmonary Parameters in Post CABG Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00712 Shafaq Wadood
Record Dates: First submitted 2020-11-03; First posted 2020-11-04 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Post-cardiac Surgery
Keywords: Ergo-meter; CABG; Endurance

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elliptical Training Group (Experimental): Total 30 minutes of elliptical cross training, including warm up, progressive elliptical training and cool down.
  Interventions: Other: Elliptical Training Group
- Ergo-metric Training Group (Experimental): Total 30 minutes of ergometric training
  Interventions: Other: Ergo-metric Training Group

INTERVENTIONS:
Other: Elliptical Training Group — The training program will be consisted of total 30 minutes of elliptical cross training (5 minutes warm up + Progressive Training up to 20 minutes of elliptical cross training + 5 minutes cool down) for 3 days in a week for 4 weeks at an average intensity of 50-70% the maximal heart rate according to ACSM guidelines.
  Arms: Elliptical Training Group
Other: Ergo-metric Training Group — The training program will be consisted of total 30 minutes of ergometric training (5 minutes warm up + Progressive Training up to 10 minutes of upper limb ergometric training + Progressive Training up to 10 minutes of lower limb ergometric training+5 minutes cool down) for 3 days in a week for 4 weeks at an average intensity of 50-70% the maximal heart rate according to ACSM guidelines.
  Arms: Ergo-metric Training Group

SUMMARY:
To determine the effects of elliptical training versus ergo-meter on cardiopulmonary parameters in post CABG patients

DETAILED DESCRIPTION:
Worldwide, physiotherapists treat patients with CAD in the acute stage following a coronary event and/ or following coronary artery bypass graft (CABG) surgery. These patients are then later followed up as outpatients during cardiac rehabilitation(CR) in turn to improve cardio-respiratory fitness and quality of life and to delay the incidence of subsequent coronary events. Early mobilisation and physical activity is often the first choice of treatment, but evidence as to the optimal intensity, timing and choice of exercises is scarce. In 2018 the effect of obesity on functional capacity, anxiety and Daily life activities in patients with coronary artery disease and phase II cardiac rehabilitation. The results shows that When Group 1 patients were assessed at the end of 30 sessions of cardiac rehabilitation (CR) program, a statistically significant improvement was detected in 6MWT, physical functioning, physical role, mental health, social functioning and pain sub parameters.

In 2019, study Changes in 6-minute walk test (6MWT) distance and heart rate walking speed index following a cardiovascular prevention and rehabilitation programme .Patients increased their 6-minute walk test distance by 40 meters and decreased their heart rate walking speed index by 2.7, which translates into a saving of three heart beats for every 100 meters walked or 45 heart beats for every mile walked.

In 2012, conducted study Resistance and Balance Training Improves Functional Capacity in Very Old Participants Attending Cardiac Rehabilitation Participants were assigned randomly in a ratio of 1:1 to an intervention group (IG; inpatient CR plus resistance training and balance training) or control group (CG;inpatient CR)after Coronary Bypass Surgery. The study concluded that there is significantly greater improvement in functional capacity measured as 6-MWD,TUG time, and maximal relative workload in the IG than in the CG..

ELIGIBILITY:
Inclusion Criteria:

* CABG patients (after 4 months) undergone phase 2 rehabilitation.

Exclusion Criteria:

* Vitally Unstable patients
* Presence of arrhythmias
* History of unstable angina in last 3 months
* Intracavitary thrombus
* Recent thrombophlebitis with or without pulmonary embolism
* Sever/e obstructive cardiomyopathies
* Uncontrolled diabetes
* Severe orthopaedic problems

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
6 min walk test: Distance (meters) | 4th week
  Changes from the baseline, 6 min walk test was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Oxygen Saturation (SpO2) | 4th week
  Changes from baseline SPO2 was measured in percentage. Oxygen immersion is the division of oxygen-soaked hemoglobin with respect to add up to hemoglobin in the blood. Pulse oximeter measure it.
Pulse Rate | 4th week
  Changes from baseline, Pulse rate was measured per minute through pulse oximeter
Modified Borg Scale of Perceived Exertion | 4th week
  Changes from the Baseline, It is a subjective numeric scale ranging from 0 to 10, where 0 indicates "no dyspnea" and 10 indicates "unbearable dyspnea." A number is chosen by the patient in order to decide the best score that matches his level of dyspnea during physical activity.
Systolic and diastolic blood pressure | 4th week
  Changes from the Baseline, Blood pressure is measured through sphygmomanometer
WHO_BREF questioner (Quality of life) | 4th week
  Changes for the baseline, The World Health Organization (WHO) Quality of Life Group Developed a self-report 26 item questionnaire called the WHO Quality of Life Instrument, Short Form (WHOQOLBREF).the questioner is intend to assess the four aspect of quality of life physical (seven questions), psychological (six questions), social (three questions), and environmental (eight questions) dimensions.There are no cut-off points above or below which quality of life could be evaluated as "poor" or "good". Thus, it was decided to rationalize the analysis by defining two groups at the extremes, both in perception of QoL and satisfaction with health (good QoL /satisfied - includes those who reported having good or very good QoL and were satisfied or very satisfied with their health; and poor QoL /dissatisfied - includes those who reported poor or very poor QoL and who were dissatisfied or very dissatisfied with their health).

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MsCPPT, Principal Investigator — Riphah International University
Locations (1):
- Rawalpindi Institute of Cardiology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ab Manap N, Khalid KBMKM, Alias MNBA, Jamaludin NB. Quality of Life among Post Acute Myocardial Infarction Patient. ILKKM Journal of Medical and Health Sciences. 2019;1(1):20-4.